### 1 Prevalence and determinants of home accidents among Turkish older men and women

#### 2 Abstract

- 3 **Background:** Home accidents are a significant public health issue in developed and developing
- 4 countries. The present study aims to identify the factors associated with home accidents among
- 5 older individuals in Türkiye.
- 6 Methods: Microdata obtained from the Türkiye Health Survey conducted by the Turkish
- 7 Statistical Institute (TUIK) in 2019 and 2022 were utilized in the present study. Binary logistic
- 8 regression analysis was used to determine factors influencing home accidents.

## 9 Results:

#### **Conclusion:**

- 11 **Keywords:** Older individuals, home accident, discrete choice model, binary logistic regression,
- 12 Türkiye

# 13

14

10

#### 1. Introduction

- Home accidents are a significant public health issue in developed and developing countries (1).
- Home refers to where older individuals spend most of their daily time, thus increasing their
- 17 likelihood of experiencing any accidents at home. Home accidents are more common among
- older individuals and can lead to serious health consequences (2). Individuals aged 65 and
- above are particularly at high risk of home accidents due to physical, psychological, and social
- 20 impairments. Musculoskeletal problems and sensory and motor function loss in this group
- 21 increase the risk of accidents (3). Home accidents are assumed to be unintentional and can range
- from minor injuries to fatalities. These accidents can occur within the home and in surrounding
- areas such as garages, gardens, terraces, and stairs (4). While unintentional home and

recreational injuries pose a risk for individuals aged 85 and older, outdoor injuries also pose a 24 risk for younger, older individuals (aged 75-79) (5). 25 26 Home accidents represent a significant health problem in terms of morbidity and mortality at older ages (6). The frequency of home accidents is found to be three times higher in women, 27 2.7 times higher in individuals living with children, 2.3 times higher in visually impaired older 28 individuals, and 2.7 times higher in older individuals with poor health status. Moreover, 29 advancing age is considered a risk factor for home accidents (7). Various home accidents 30 31 include falls, burns, crushes, cuts, and electric shocks (8). Around 80% of injuries that necessitate medical attention take place within the home environment, with a significant portion 32 of these injuries, approximately two-thirds, being classified as serious injuries, predominantly 33 34 resulting from falls and burns (5). 35 Similar to the global trend, the older population in Türkiye is rapidly increasing (9). While the global average older population ratio was 9.9% in 2022, Türkiye's older population ratio of 36 9.8% is close to the global average (10). These data indicate that Türkiye has a significantly 37 more ageing population (11). The prevalence of older individuals experiencing at least one 38 accident in Türkiye is 38.6%, with falls being the most common accident at 63.3% (6). As 39 reported in another study, more than half of the older population had experienced a home 40 accident in the previous year (59.4%), with falls (70.2%) and kitchen accidents (31.7%) ranking 41 42 at the top (12). Epidemiological characteristics of injured patients were examined in Tehran, 43 where traffic accidents and falls were identified as the two most common causes of injury (13). 44 Falls in the home environment account for over 33% of accidents and are the second leading cause of death and the main cause of injury in more than 41.2% of cases. Falls during patient 45 admissions also impose additional burdens and costs on the healthcare system (14). The total 46 medical cost for treating fatal and non-fatal fall injuries in older adults exceeded \$50 billion in 47 the USA in 2015 (15). "Falls" occurring in the bathroom, hallway, living room, or bedroom,

48

originating from the floor or stairs, can result in doctor visits and hospitalizations (1). Factors contributing to increased home injuries include advanced age, economic hardships, obesity, and comorbidities (5). Among older adults living in the community, a significant proportion of falls, ranging from 10% to 38%, lead to non-fatal injuries, hospitalizations, disability, or a decline in independence (16-18). Various risk factors have been identified in association with falls, including advanced age, a history of previous falls, muscle weakness, difficulties with walking and balance, dementia, impaired vision, arthrosis, diabetes, stroke, Parkinson's disease, and urinary incontinence (19). Burns constitute another type of home accident in older individuals. Burn injury is one of the most devastating types of trauma affecting millions of people worldwide, leading to severe morbidity and mortality, with individuals aged 65 and above being the most affected demographic group. The presence of comorbidities in older individuals leads to higher morbidity and mortality in burns due to age-related changes in the central and peripheral nervous system (20). Older individuals may also experience traumas as a result of accidents that occur within their homes. These traumas can have severe consequences for older adults, leading to increased rates of illness and death (21). The proportion of older individuals presenting to Level I and II trauma centers was 23% in 2003, which increased to 30% in 2009 (22). This rate is expected to reach 39% by 2050 (23). The cost of home accidents is estimated to be 3.5 times higher than that of traffic accidents (24). Decreased capacities of older individuals often result in limitations in daily life activities. Ageing and declining individual capacities increase the prevalence of disease and disability among older individuals. Living at home, associated with independence and autonomy-related physical, psychological, and psychosocial benefits, is a desired and essential goal for older individuals (25). Therefore, it is necessary to examine the factors contributing to home

49

50

51

52

53

54

55

56

57

58

59

60

61

62

63

64

65

66

67

68

69

70

71

72

73

- accidents among older individuals to ensure home safety. Hence, this study investigates the risk
- 75 factors affecting home accidents among older individuals in Türkiye.

#### **2. Method**

- 77 This section will explain the specifics of the data utilized in the research, the variables
- categorized as dependent and independent, and the methodology employed in the study.

### 79 **2.1. Data**

- 80 The research utilised microdata from the Türkiye Health Survey, published by the Turkish
- Statistical Institute (TUIK) in 2019 and 2022. The most recent data available from TUIK's
- 82 health survey is 2022. The Türkiye Health Survey is a significant research endeavour that
- 83 reflects the entire country and enables national and international comparisons. The dataset
- offers a wide range of health indicators related to the well-being of infants, children, and adults,
- along with insights into individuals' access to healthcare services (26).

# 2.2. Outcome Variables

- 87 Older individuals are at risk for home accidents due to their developmental characteristics (2,
- 88 3).

86

94

- 89 The data obtained from individuals aged 60 and above were used in this study. The study's
- 90 dependent variable is the occurrence of home accidents, measured by the question, "Have you
- 91 experienced a home accident resulting in injury in the last 12 months? (Yes, No)." In the
- 92 established model, the dependent variable categories are assigned 1 if the individual has
- experienced a home accident and 0 if they have not.

# 2.3. Independent variables

- The independent variables included in the study are those available in the Türkiye Health
- 96 Survey. These variables were selected as risk factors based on the literature (5, 7, 19, 27-33).

The independent variables of this study are gender (female, male), education level (illiterate/less than primary school, primary school, secondary school and above), marital status (single, married), employment status (unemployed, employed), general health status (very good/good, fair, poor/very poor), presence of arthrosis (no, yes), urinary incontinence (no, yes), wearing glasses (yes/cannot see at all, no), experiencing difficulty in carrying or holding items (no difficulty, some difficulty/considerable difficulty/cannot do at all), experiencing difficulty in affording health care services (no, yes), and survey year (2019, 2022).

# 2.4. Statistical Analysis

Survey statistics in Stata 15 (Stata Corporation) were utilized to address the complex sampling design and weights. Weighted analysis was conducted. Initially, frequencies and percentages were obtained considering the home accident occurrence and years among the older participants. Then, binary logistic regression analyses were employed to identify the risk factors influencing home accidents in older individuals.

### 3. Results